CLINICAL TRIAL: NCT01068925
Title: An Open-Label, Single Sequence, Three-Period Drug Interaction Study of GSK1349572 and Tipranavir/Ritonavir in Healthy Adult Subjects (ING113096)
Brief Title: Drug Interaction Study Between GSK1349572 and Tipranavir/Ritonavir in Healthy Volunteers
Acronym: ING
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 113096
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: healthy volunteer; pharmacokinetics; HIV, GSK1349572, tipranavir, ritonavir, drug interaction
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARM 1 (Experimental): Arm 1:
  GSK1349572 QD for 5 days (Treatment A).
  Interventions: Drug: GSK1349572
- ARM 2 (Experimental): ARM 2: TPV/RTV 500/200mg BID (Treatment B).
  Interventions: Drug: GSK1349572
- ARM 3 (Experimental): ARM 3: GSK1349572 50mg QD and TPV/RTV 500/200mg BID (Treatment C).
  Interventions: Drug: GSK1349572

INTERVENTIONS:
Drug: GSK1349572 — 1. GSK1349572 QD x 5 days
  2. TPV/RTV 500/200mg BID x 7 days
  3. GSK1349572 50mg QD and TPV/RTV 500/200mg BID x 5 days
  Other Names: TPV/RTV 500/200mg BID x 7 days; GSK1349572 QD x 5 days; GSK1349572 50mg QD and TPV/RTV 500/200mg BID x 5 days

SUMMARY:
The purpose of this study is to determine whether there is a drug interaction between GSK1349572 and the HIV protease inhibitors Tipranavir/Ritonavir (TPV/RTV).

DETAILED DESCRIPTION:
The construction of a new antiretroviral regimen with GSK1349572 in raltegravir-resistant subjects will likely require less commonly used agents such as tipranavir and enfuvirtide. Ritonavir-boosted tipranavir (TPV/RTV) has been shown to induce drug metabolizing enzymes and lead to decreased exposure of some antiretrovirals thus necessitating a drug interaction study with GSK1349572 as GSK1349572 is eliminated primarily by metabolism.

This is a single-center, single sequence, open-label, three-period study, in adult male and female healthy subjects. Approximately 18 subjects will receive GSK1349572 50mg QD for 5 days (Treatment A). Subjects will then be administered TPV/RTV 500/200mg BID for 7 days (Treatment B) followed by the combination of GSK1349572 50mg QD and TPV/RTV 500/200mg for 5 days (Treatment C). There will be no washout periods between treatments. Safety evaluations will be collected during each treatment period. Serial PK samples for GSK1349572 will be collected and compared between Treatment A and C. A follow-up visit will occur 7-14 days after the last dose of study drug.

The study will be conducted at one centre in the US with healthy adult male and female subjects.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply: (a single repeat is allowed for assessments to determine eligibility).

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* AST, ALT, alkaline phosphatase and bilirubin within normal ranges. A single repeat is allowed to determine eligibility.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy or bilateral oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to continue to use contraception until at least 3 days after the last dose of study drug.
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women and body mass index (BMI) within the range 18.5 -31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, including sulfa-containing drugs, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, antacids, iron supplements, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Use of NSAIDs or aspirin compounds within 21 days of the first dose of study medication.
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* History of regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
* Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* Any patient with a history of bleeding diathesis, gastrointestinal bleeding or at increased risk of bleeding such as frequent nose bleeds, high blood pressure, heavy menses, von Willebrand disease, and personal or family history of bleeding disorders
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* History of significant renal or hepatobiliary diseases.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of 2nd degree or higher AV block.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination):

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02-15 (Actual); Primary Completion 2010-04-05 (Actual); Study Completion 2010-04-05 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1349572 steady-state AUC(0-tau), Cmax, C0, Ctau, and Cmin following administration of GSK1349572 50mg QD for 5 days and following co-administration with TPV/RTV 500/200mg BID for 5 days. | 17 days

SECONDARY OUTCOMES:
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, ECG, and vital signs assessments. | 31 days
Plasma GSK1349572 PK parameters: tmax, tmin, CL/F and t½, following administration of GSK1349572 50mg QD for 5 days and following co-administration with TPV/RTV 500/200mg BID for 5 days | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- [Background] Song I, Borland J, Chen S, Guta P, Lou Y, Wilfret D, Wajima T, Savina P, Peppercorn A, Castellino S, Wagner D, Hosking L, Mosteller M, Rubio JP, Piscitelli SC. Effects of enzyme inducers efavirenz and tipranavir/ritonavir on the pharmacokinetics of the HIV integrase inhibitor dolutegravir. Eur J Clin Pharmacol. 2014 Oct;70(10):1173-9. doi: 10.1007/s00228-014-1732-8. Epub 2014 Aug 23. PMID 25146692